CLINICAL TRIAL: NCT07335796
Title: A Phase 2 Study of Androgen Deprivation Therapy and BMS986365 in High-Risk Localized Prostate Cancer Patients Prior to Radical Prostatectomy
Brief Title: A Study of BMS986365 in Combination With Degarelix in People With Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-262
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Memorial Sloan Kettering Cancer Center; 25-262
MeSH Terms: conditions — Prostatic Neoplasms | interventions — deucravacitinib; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with high-risk localized prostate cancer (Experimental): Eligible participants with high-risk localized prostate cancer based on one or more of the following: PSA >20ng/ml, Gleason Score ≥8, or Clinical stage ≥cT3a.
  Interventions: Drug: BMS-986165; Drug: Degarelix

INTERVENTIONS:
Drug: BMS-986165 — BMS986365 (CC-94676) is an androgen receptor (AR) ligand-directed degrader that was designed to target the AR for degradation in castration-resistant prostate cancer (CRPC)
Drug: Degarelix — Degarelix is a GnRH antagonist that blocks the action of GnRH on the pituitary and effectively suppresses testosterone production

SUMMARY:
The purpose of this study is to find out whether BMS986365 in combination with degarelix, given before standard surgical treatment (radical prostatectomy), is a safe and effective treatment that causes few or mild side effects for people who have localized high-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant or participant's legally authorized representative (LAR) is willing and able to provide written informed consent and privacy authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.
* Individuals with prostate cancer 18 years of age and above
* Histological or cytological evidence of prostate cancer
* Documented high-risk localized prostate cancer based on one or more of the following NCCN criteria:

  1. PSA ≥ 20ng/ml or
  2. Gleason ≥8 or
  3. Clinical stage ≥cT3a
* Candidate for RP as determined by treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal organ function with acceptable initial laboratory values within 28 days of registration:

ANC ≥ 1.5 K/mcL Hemoglobin ≥ 9g/dL Platelet count ≥ 100 K/mcL Potassium* within institutional normal range Calcium* within institutional normal range Magnesium* within institutional normal range Total Bilirubin ≤ 1.5 x ULN (Note: In participants with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, participant may be eligible) SGOT (AST) ≤ 2.5 x ULN SGPT (ALT) ≤ 2.5 x ULN CrCl** > 60 mL/min *If these electrolytes are corrected with supplements, eligibility should be confirmed prior to the first dose of study intervention.

**Using Cockcroft-Gault equation or measured CrCl using 24-hour urine collection

- Male Participants: i) A participant who is sexually active with individuals of childbearing potential (IOCBP) must agree to follow instructions for method(s) of contraception as described below and included in the informed consent form.

Note: Azoospermic males are not exempt from contraceptive requirements and will be required to always use a latex or other synthetic condom during any sexual activity (e.g., vaginal, anal, oral) with IOCBP, even if the participant has undergone a successful vasectomy or if the partner is pregnant. ii) Participants will be required to always use a latex or other synthetic condom during any sexual activity (e.g., vaginal, anal, oral) with IOCBP, even if the participant has undergone a successful vasectomy or if the partner is pregnant or breastfeeding. Male (as assigned at birth) participants should continue to use a condom during the intervention period and for at least 2 months (for BMS-986365) and as per the label for degarelix after the last dose of study intervention.

iii) IOCBP partners of participants should be advised to use a highly effective method of contraception during the intervention period and for at least 2 months (for BMS-986365) and as per the label for degarelix after the last dose of study intervention for the male participant.

iv) Participants with a pregnant or breastfeeding partner must agree to remain abstinent from sexual activity or use a male condom during any sexual activity (eg, vaginal, anal, oral), even if the participant has undergone a successful vasectomy, during the intervention period and for at least 2 months (for BMS-986365) and as per the label for degarelix after the last dose of study intervention. v) Participants must refrain from donating sperm during the intervention period and for at least 2 months (for BMS-986365) and as per the label for degarelix after the last dose of study intervention. vi) Breastfeeding partners of participants should be advised to consult their health care provider about using appropriate highly effective contraception during the time the male participant is required to use condoms.

See Appendix B for further guidelines and definitions.

Exclusion Criteria:

* Radiographic evidence of distant (extra-pelvic) metastatic prostate cancer on CT and/or MRI, bone scan or PET scan (any PET modality)

Patients with N1 disease may be eligible for the study if planned for a radical prostatectomy per standard-of-care/institutional guidelines.

* On ADT (GnRH agonists or antagonists) for > 4 weeks at time of consent
* Other than ADT as mentioned in 6.2.2, prior systemic therapy for treatment of their prostate cancer, including but not limited to chemotherapy, immunotherapy, etc.
* Prior local therapy to the prostate for prostate cancer, including but not limited to radiation, HIFU, phototherapy, etc.
* Participants who are considered a poor medical risk due to a serious, uncontrolled medical disorder, or recovering from a recent surgery (approximately within 1 month, or as deemed recent per surgeon), for which in the opinion of the investigator would interfere with treatment on this study.
* Any patient who cannot swallow oral medications or have gastrointestinal disorders in the opinion of the investigator are likely to interfere with absorption.
* Participant has impaired cardiac function or clinically significant cardiac disease, including any of the following:

  i. LVEF < 50% as determined by ECHO or MUGA scan at Screening. ii. Complete left bundle branch, high-grade AV block (eg, bifascicular block, Mobitz type II and third-degree AV block), or other clinically significant abnormal ECG finding at Screening. Participant with a permanent pacemaker are excluded. iii. History of clinically significant sinus bradycardia or sick sinus syndrome or bradycardia with heart rate < 50 bpm at Screening. (Note: All is determined by the average of the triplicate Screening ECG, based on local reading.)
  1. A prolongation of the QT interval on Screening ECG as defined by repeated demonstration of a QTc interval ≥ 450 ms using QTcF.
  2. Participant would be excluded if the QTcF interval cannot be determined on the Screening ECG (eg, unreadable or not interpretable).
  3. In the presence of right bundle branch block, if measured QTcF is > 450 ms at baseline, then the ECG for QTc reading should be verified by a cardiologist to confirm eligibility. iv. A history of sustained ventricular tachycardia, ventricular fibrillation, TdP, or resuscitated cardiac arrest, individual or family history of long QT syndrome, or cardiomyopathy. v. Concurrent treatment with antiarrhythmic or other drugs that prolong the QT interval.

     For study eligibility, a washout period of ≥ 5 half-lives must have elapsed prior to the first dose of study intervention. vi. Congestive heart failure (New York Heart Association Class III or IV) ≤ 12 months prior to the first dose of study intervention. vii. Myocardial infarction, myocarditis, or pericarditis ≤ 6 months prior to the first dose of study intervention. viii. Unstable or poorly controlled angina pectoris (including the Prinzmetal variant of angina pectoris) or symptomatic peripheral vascular disease. ix. Poorly controlled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg).

     Participants with a history of hypertension can be enrolled if the investigator considers that BP is controlled by antihypertensive treatment.
* Participants with clinically significant venous thromboembolism (eg, pulmonary embolism and deep vein thrombosis) within 3 months prior to the first dose of study intervention.
* Active viral hepatitis, including the following:

  i. Any positive test result for HBV indicating presence of virus, eg, HBV DNA positive would be excluded. Participants with anti-HBs positive in line with prior vaccination are eligible to enroll. ii. Any positive test result for HCV indicating presence of active viral replication (detectable HCV-RNA). iii. Participants with positive HCV antibody and an undetectable HCV RNA are eligible to enroll.
* Known HIV positive with an AIDS defining opportunistic infection within the last year, or a current CD4 count < 350 cells/μL. Participants with HIV are eligible if: i. Participant has received ART for at least 4 weeks prior to treatment assignment as clinically indicated while enrolled on study and an HIV viral load less than 400 copies/mL prior to enrollment. ii. Participant continues on ART as clinically indicated while enrolled on study.

iii. In the case ART is at risk of drug-drug interaction, participants should be switched to an alternate effective ART regimen (with minimal drug-drug interaction potential) before study participation or should be excluded from the study if their regimen cannot be altered. iv. CD4 counts and viral load are monitored per standard of care by a local health care provider.

* Any other active malignancy at time of first dose of study treatment or diagnosis of another malignancy within 3 years prior to first dose of study treatment that requires active treatment, except for basal or squamous cell skin cancer or superficial bladder cancer that has previously been treated.
* Use of any prohibited concomitant medications including herbal supplements (Section 10.4) within 2 weeks prior to treatment start
* Receiving any other investigational agents within 4 weeks or 5x the half-life of investigational agent (whichever is longer) from this study's treatment start
* Known allergy to any of the compounds under investigation
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2030-01-09 (Estimated); Study Completion 2030-01-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of pathologic complete response/pCR | 42 months
  The primary objective is to determine the frequency of achieving a pathologic complete response (pCR) and/or minimal residual disease (MRD defined as ≤ 5 mm tumor) .

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Lacuna, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made following one year after publication and for up to 36 months later. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org